CLINICAL TRIAL: NCT02301338
Title: Improving Health of Patients With Colon Cancer Following Surgery: A Trial of SA-ICAN Via Videoconferencing
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-213
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Colon Cancer
Keywords: Videoconferencing; Following Surgery; 14-213
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Usual Care: The patient will get instructions on: - Follow-up appointment date/time with your surgeon - Proper diet - Medications - Communicating concerning symptoms with the surgeon
  The patient will answer questions on:
  * Social support
  * Quality of life
  Interventions: Other: Usual care
- Phone Calls: In addition to what the usual care group gets, the patient will also receive weekly phone calls by a geriatrics RN following hospital discharge.
  The patient will answer questions on:
  * Social support
  * Quality of life
  Interventions: Other: Usual care; Other: Phone Calls

INTERVENTIONS:
Other: Usual care
Other: Phone Calls
  Groups: Phone Calls

SUMMARY:
The purpose of this study is to assess the impact of more frequent follow-up (by videoconference) of these patients. Videoconference is a method of communication over a distance. In this method, the patient will hear the person's voice (like on the telephone) and will see that person over video.

The study will compare more frequent follow-up of patients by videoconferencing to routine follow-up of patients. The investigators will compare each type of follow-up to see the effect on the number of times patients need to visit emergency rooms or need admission to hospitals. The study will also look at the difference between each type of follow-up on patients' quality of life and social support thirty days after hospital discharge.

The study will also measure satisfaction and acceptability of this intervention among those who had follow-ups by videoconference.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older.
* Newly diagnosed cancer.
* Referred to the geriatrics service for pre-operative evaluation before surgical resection of his/her tumor.

Exclusion Criteria:

* Inability to comprehend English.
* Deafness , measured by the Hearing Handicap Inventory for the Elderly Screening Version (HHIE-S) [16], score equal or above 30. (appendix 5)
* Cognitive impairment (score of 0-1 in Mini-Cog Test).
* Nursing home resident.
* Planned hospital length of stay of one day or less.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Newly diagnosed older colon cancer patients require pre-operative evaluation before undergoing surgery.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
acute healthcare utilization (AHCU) rates | 30 days post -discharge
  (i.e. hospital readmission and/or ER visit)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Shahrokni, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/